CLINICAL TRIAL: NCT03383367
Title: Extending the Prerogatives of Colorectal Cancer Screening French Organizations to the Follow-up After Colonoscopy of Patients Aged 50 or More: Pilot Study in the Rhône Administrative Department
Brief Title: Colorectal Cancer Screening French Organizations for the Follow-up After Colonoscopy
Acronym: Tempo-colo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Association pour le Dépistage Organisé des Cancers dans le Rhône (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2016-A01710-51
Record Dates: First submitted 2017-12-01; First posted 2017-12-26 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Colorectal Cancer
Keywords: mass screening; colonoscopy surveillance; high risk patients
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: A prospective interventional study to evaluate the impact of a reminder sent by the Adémas-69 organization to improve coloscopy surveillance and compliance with recommendations for high risk of colorectal cancer people.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tempo Colo (Experimental)
  Interventions: Behavioral: Tempo Colo

INTERVENTIONS:
Behavioral: Tempo Colo — Reminder letter for people at high risk of colorectal cancer.

SUMMARY:
France is one of the European countries where the incidence of colorectal cancer is the highest among cancers for both sexes. Fecal occult blood screening has been implemented since 2008. However, this screening excludes high risk people who have a 10 to 30 % risk of developing a CRC during their lifetime. Colonoscopy follow up of these persons is not organized, and it is up to the attending physician to recall the date of the surveillance colonoscopy. This results in a poor compliance with the recommendations by these people. A postal reminder of the surveillance colonoscopies sent by The French screening organizations to the patients should increase adherence to follow-up recommendations. The colorectal cancer screening organizations will collects from the hepatogastroenterologists (HGE) informations on colonoscopies of people more than 50 years old who live in the Rhone. These informations will allow to send a reminder 3 months before the date recommended by the HGE. Participation rate and timeliness will be assessed, as well as the severity of the lesions found. A medico-economic analysis will also be carried out.

ELIGIBILITY:
Inclusion Criteria:

* people aged 50 years or more ;
* at high risk of colorectal cancer ;
* living in Rhône administrative departement or Metropolitan Lyon

Exclusion Criteria:

* person with chronic inflammatory bowel disease
* colorectal cancer in diagnosis or treatment period

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33000 (Estimated)
Dates: Start 2017-08-24 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
participation rate at future colonoscopy | At time of evaluation we will check the colonoscopy realized at six months after sending the letter at the person
  participation rate at future colonoscopy that is the number of patient that really have colonoscopy among the patients who receive a reminder letter The systematic registry of colonoscopies will permit to assess if a patient performs it.

SECONDARY OUTCOMES:
description of lesions severities found at surveillance colonoscopy after letter reminder | Lesions'severity will be evaluated at 6, 9 or 15 months following the reminder sent according to the colonoscopist's recommendation (1,3 or 5 years after reference exams). By the way of systematic registration. .
  We will assess the severity of the lesions found at colonoscopy performed at th right time : level of dysplasia ; size ; histologic characteristics ; numbers of adenoma.
Cost-utility analysis of the reminder letter for surveillance colonoscopy | Lesions'severity will be evaluated at 6, 9 or 15 months following the reminder sent according to the colonoscopist's recommendation (1,3 or 5 years after reference exams). The costs will be registered at the same time.
  French Health Insurance is the point of vue selected for the evaluation. It's a cost-utility analysis. A Markov model will be performed. The data will proceed from litterature and from data registration during the study. A complementary study will be performed specifically if needed.
  For the Markov model the data needed : neoplasia, adenocarcinoma, advanced adenoma, reminders costs, treatments costs, examinations costs, organization costs.

CONTACTS AND LOCATIONS:
Locations (1):
- Adémas-69, Lyon, Rhône, France